CLINICAL TRIAL: NCT00067769
Title: Treatment of Early Childhood Constipation/Encopresis
Brief Title: Internet-based Treatment of Early Childhood Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, Department of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11116; 5R01HD028160-12 (NIH)
Record Dates: First submitted 2003-08-27; First posted 2003-08-28 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2014-06

CONDITIONS: Encopresis
Keywords: Encopresis; Internet; Web; Treatment; Intervention
MeSH Terms: conditions — Encopresis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU (Active Comparator): Patients received treatment as usual (TAU) as defined as continued clinical care.
  Interventions: Behavioral: treatment as usual
- TAU+UCanPoopToo (Experimental): Patients received treatment as usual (TAU) plus the Internet intervention (UCanPoopToo.)
  Interventions: Behavioral: Internet-based intervention UCanPoopToo

INTERVENTIONS:
Behavioral: Internet-based intervention UCanPoopToo — Internet-based intervention to administer Enhanced Toilet Training (ETT).
  Arms: TAU+UCanPoopToo
Behavioral: treatment as usual — Routine clinical care.
  Arms: TAU

SUMMARY:
Encopresis, also known as fecal incontinence, is the voluntary or involuntary passage of stools causing soiling of clothes by a child over 4 years of age. The purpose of this study is to evaluate an Internet intervention for the treatment of encopresis.

DETAILED DESCRIPTION:
An estimated 2.3% of children suffer from encopresis. Enhanced Toilet Training (ETT) is one of the most effective ways of treating this disorder. When delivered by skilled and knowledgeable clinicians, ETT is twice as effective as intensive medical management alone. Although ETT is effective in treating encopretic children, there are six major barriers to its implementation: 1) availability of a knowledgeable and skilled clinician; 2) parental acceptance of referral to a mental health professional; 3) expense of service; 4) burden of time and distance to access such specialty services; 5) child resistance to disclosure of embarrassing material; and 6) willingness of the child and parent to follow treatment recommendations. This project will circumvent these barriers by developing an interactive Internet-based ETT program. The study will then assess the feasibility of the program by determining the acceptance, function, and effectiveness of the intervention.

This project will have four phases. Phase 1 will identify optimal Internet and treatment elements as well as issues in need of experimental investigation. Phase 2 will investigate how to enhance Internet interventions. Phase 3 will evaluate the relative benefit of adding the Internet treatment to clinical services provided by clinicians in the fields of medicine and mental health. Phase 4 will investigate the relative long-term benefits of adding such an Internet-based intervention to professional care to determine its impact on symptom improvement, relapse prevention, quality of life, and its cost-effectiveness. Phase 4 will also assess to what extent the program is disseminated worldwide when made available on the Internet.

ELIGIBILITY:
Inclusion Criteria

* Child seen by pediatrician, family physician, or psychologist for the treatment of encopresis
* Access to the Internet, either through a family computer or a community computer

Exclusion Criteria

* Diagnosis of either mental retardation (IQ < 85) or
* A primary illness responsible for fecal soiling (e.g., spina bifida)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2003-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Fecal accident outcomes with online diary data | Pre, Post (4-6 weeks), and one year Post after the intervention period (4-6 weeks)
  Number of accidents per 2 week period
Success and cure rates | Post (4-6 weeks) and one year Post after the intervention period (4-6 weeks)
  Success rate as defined by having zero or one fecal accident over a two week period. Cure rate as defined by having zero accidents over the previous two weeks.

SECONDARY OUTCOMES:
Fecal accident outcomes with retrospective data | Pre, Post (4-6 weeks), and one year Post after the intervention period (4-6 weeks)
  Number of accidents per 2 week period
Parent knowledge of encopresis | Pre, Post (4-6 weeks), and one year Post after the intervention period (4-6 weeks)
  Parent knowledge of encopresis was assessed on a revised version of the Encopresis Knowledge Scale (EKS).
Virginia Encopresis Constipation Apperception Test (VECAT) | Pre, Post (4-6 weeks), and one year Post after the intervention period (4-6 weeks)
  Parent assessment of child's bowel specific problems related to encopresis and constipation.
Encopresis Cost Analysis | Pre and Post (4-6 weeks)
  Participants quantified items and events that occurred which contribute to the cost of encopresis such as number of diapers used, number of school days missed, number of parent trips to school, and clean-out procedures then cost estimates were applied to each.

OTHER OUTCOMES:
Usage patterns of the Internet intervention | Post (4-6 weeks)
  Usage (number of Cores completed; number of Follow-ups completed and Modules assigned)
Internet Intervention Utility Measure of Satisfaction | Post (4-6 weeks)
  Parent and child rated their satisfaction with the Internet intervention using the Internet Intervention Utility Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Ritterband LM, Cox DJ, Walker LS, Kovatchev B, McKnight L, Patel K, Borowitz S, Sutphen J. An Internet intervention as adjunctive therapy for pediatric encopresis. J Consult Clin Psychol. 2003 Oct;71(5):910-7. doi: 10.1037/0022-006X.71.5.910. PMID 14516239
- [Background] Cox DJ, Morris JB Jr, Borowitz SM, Sutphen JL. Psychological differences between children with and without chronic encopresis. J Pediatr Psychol. 2002 Oct-Nov;27(7):585-91. doi: 10.1093/jpepsy/27.7.585. PMID 12228330
- [Background] Borowitz SM, Cox DJ, Sutphen JL, Kovatchev B. Treatment of childhood encopresis: a randomized trial comparing three treatment protocols. J Pediatr Gastroenterol Nutr. 2002 Apr;34(4):378-84. doi: 10.1097/00005176-200204000-00012. PMID 11930093
- [Background] Brooks RC, Copen RM, Cox DJ, Morris J, Borowitz S, Sutphen J. Review of the treatment literature for encopresis, functional constipation, and stool-toileting refusal. Ann Behav Med. 2000 Summer;22(3):260-7. doi: 10.1007/BF02895121. PMID 11211851
- [Background] Borowitz SM, Cox DJ, Sutphen JL. Differences in toileting habits between children with chronic encopresis, asymptomatic siblings, and asymptomatic nonsiblings. J Dev Behav Pediatr. 1999 Jun;20(3):145-9. doi: 10.1097/00004703-199906000-00002. PMID 10393070
- [Background] Cox DJ, Sutphen J, Borowitz S, Kovatchev B, Ling W. Contribution of behavior therapy and biofeedback to laxative therapy in the treatment of pediatric encopresis. Ann Behav Med. 1998 Spring;20(2):70-6. doi: 10.1007/BF02884451. PMID 9989311
- [Background] Cox DJ, Sutphen J, Ling W, Quillian W, Borowitz S. Additive benefits of laxative, toilet training, and biofeedback therapies in the treatment of pediatric encopresis. J Pediatr Psychol. 1996 Oct;21(5):659-70. doi: 10.1093/jpepsy/21.5.659. PMID 8936895
- [Background] Ling W, Cox DJ, Sutphen J, Borowitz S. Psychological factors in encopresis: comparison of patients to nonsymptomatic siblings. Clin Pediatr (Phila). 1996 Aug;35(8):427. doi: 10.1177/000992289603500814. No abstract available. PMID 8862907